CLINICAL TRIAL: NCT00925301
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Pharmacodynamics of AT1001 in Patients With Fabry Disease and AT1001-Responsive GLA Mutations
Brief Title: Study of the Effects of Oral AT1001 (Migalastat Hydrochloride) in Patients With Fabry Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AT1001-011; FACETS (Other: Amicus Therapeutics); 2009-013459-31 (EudraCT Number)
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Fabry Disease
Keywords: Amicus Therapeutics; AT1001; Migalastat; Pharmacokinetics; Substrate; Galafold
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor and Assessor were also blinded
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Migalastat (Experimental): Migalastat 150-mg capsule taken orally every other day (QOD) for 6 months and an open-label 6-month treatment extension, followed by an optional, 12-month, open-label treatment extension.
  Interventions: Drug: migalastat hydrochloride
- Placebo (Placebo Comparator): Placebo capsule taken orally QOD for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: migalastat hydrochloride — Oral capsule QOD
  Other Names: AT1001; Galafold; Migalastat
  Arms: Migalastat
Drug: Placebo — Oral capsule QOD
  Arms: Placebo

SUMMARY:
The primary objective of this study was to compare the effect of migalastat (123 milligrams [mg] of migalastat [equivalent to 150 mg of migalastat hydrochloride]) (migalastat) versus placebo on kidney globotriaosylceramide (GL-3).

DETAILED DESCRIPTION:
This double-blind, randomized, placebo-controlled study was conducted in 67 participants at 46 sites worldwide. The study consisted of 2 stages and an optional open-label treatment extension phase:

Stage 1 included a screening period of up to 2 months followed by a 6-month treatment period which involved 4 visits to the clinic. Participants were randomized in equal proportions to receive either migalastat or placebo.

After completing the 6-month double-blind phase, all participants entered Stage 2 of the study and received migalastat in an open-label manner. Stage 2 treatment lasted for 6 months and involved up to 4 visits to the clinic.

Participants who completed both Stage 1 and Stage 2 of the study as scheduled were offered the opportunity to participate in an open-label treatment extension phase with migalastat. The open-label treatment extension phase lasted 12 months and involved 2 visits to the clinic. A follow-up visit was undertaken 1 month following completion or discontinuation from the open-label treatment extension. Participants completing the 12-month open-label treatment extension and providing consent to enter a separate long-term extension were not required to complete this follow-up visit.

Study assessments included clinical laboratory tests, 12-lead electrocardiogram, kidney biopsy, kidney function testing, echocardiography, and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 16 and 74 diagnosed with Fabry disease.
* Confirmed mutant form of α-galactosidase A shown to be responsive to migalastat in vitro.
* Participant has never been treated with enzyme replacement therapy (ERT) or has not received ERT for 6 consecutive months or longer before the screening visit for the study.
* Urine GL-3 ≥4 times the upper limit of normal at screening.
* Participants taking angiotensin converting enzyme inhibitors or angiotensin receptor blockers must be on a stable dose for a minimum of 4 weeks before the baseline visit.
* Females who can become pregnant and all males agree to be sexually abstinent or use medically accepted methods of birth control during the study and for 30 days after study completion.
* Participant is willing and able to provide written informed consent and assent, if applicable.

Exclusion Criteria:

* Participant has undergone or is scheduled to undergo kidney transplantation, or is currently on dialysis.
* Estimated glomerular filtration rate <30 milliliters per minute per 1.73 meters squared (chronic kidney disease Stage 4 or 5) based on the Modification of Diet in Renal Disease equation at screening.
* Pregnant or breast-feeding.
* History of allergy or sensitivity to study medication (including excipients) or other iminosugars (for example, miglustat, miglitol).
* Participant is treated or has been treated with any investigational drug within 30 days of study start.
* Participant is currently treated or has ever been treated with migalastat.

Ages: 16 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-10-23 (Actual); Primary Completion 2012-06-12 (Actual); Study Completion 2014-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (28):
- United States (13):
  - Los Angeles, California
  - San Francisco, California
  - Decatur, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - New York, New York
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Salt Lake City, Utah
  - Springfield, Virginia
  - Seattle, Washington
- Buenos Aires, Argentina
- Australia (2):
  - Adelaide
  - Parkville
- Brazil (2):
  - Porto Alegre
  - São Paulo
- Montreal, Quebec, Canada
- Copenhagen, Denmark
- Cairo, Egypt
- Garches, France
- Roma, Italy
- Warsaw, Poland
- Spain (2):
  - Barcelona
  - Zaragoza
- Ankara, Turkey (Türkiye)
- Salford, United Kingdom

REFERENCES:
- [Derived] Bichet DG, Aerts JM, Auray-Blais C, Maruyama H, Mehta AB, Skuban N, Krusinska E, Schiffmann R. Assessment of plasma lyso-Gb3 for clinical monitoring of treatment response in migalastat-treated patients with Fabry disease. Genet Med. 2021 Jan;23(1):192-201. doi: 10.1038/s41436-020-00968-z. Epub 2020 Sep 30. PMID 32994552
- [Derived] Germain DP, Nicholls K, Giugliani R, Bichet DG, Hughes DA, Barisoni LM, Colvin RB, Jennette JC, Skuban N, Castelli JP, Benjamin E, Barth JA, Viereck C. Efficacy of the pharmacologic chaperone migalastat in a subset of male patients with the classic phenotype of Fabry disease and migalastat-amenable variants: data from the phase 3 randomized, multicenter, double-blind clinical trial and extension study. Genet Med. 2019 Sep;21(9):1987-1997. doi: 10.1038/s41436-019-0451-z. Epub 2019 Feb 6. PMID 30723321
- [Derived] Schiffmann R, Bichet DG, Jovanovic A, Hughes DA, Giugliani R, Feldt-Rasmussen U, Shankar SP, Barisoni L, Colvin RB, Jennette JC, Holdbrook F, Mulberg A, Castelli JP, Skuban N, Barth JA, Nicholls K. Migalastat improves diarrhea in patients with Fabry disease: clinical-biomarker correlations from the phase 3 FACETS trial. Orphanet J Rare Dis. 2018 Apr 27;13(1):68. doi: 10.1186/s13023-018-0813-7. PMID 29703262
- [Derived] Benjamin ER, Della Valle MC, Wu X, Katz E, Pruthi F, Bond S, Bronfin B, Williams H, Yu J, Bichet DG, Germain DP, Giugliani R, Hughes D, Schiffmann R, Wilcox WR, Desnick RJ, Kirk J, Barth J, Barlow C, Valenzano KJ, Castelli J, Lockhart DJ. The validation of pharmacogenetics for the identification of Fabry patients to be treated with migalastat. Genet Med. 2017 Apr;19(4):430-438. doi: 10.1038/gim.2016.122. Epub 2016 Sep 22. PMID 27657681
- [Derived] Germain DP, Hughes DA, Nicholls K, Bichet DG, Giugliani R, Wilcox WR, Feliciani C, Shankar SP, Ezgu F, Amartino H, Bratkovic D, Feldt-Rasmussen U, Nedd K, Sharaf El Din U, Lourenco CM, Banikazemi M, Charrow J, Dasouki M, Finegold D, Giraldo P, Goker-Alpan O, Longo N, Scott CR, Torra R, Tuffaha A, Jovanovic A, Waldek S, Packman S, Ludington E, Viereck C, Kirk J, Yu J, Benjamin ER, Johnson F, Lockhart DJ, Skuban N, Castelli J, Barth J, Barlow C, Schiffmann R. Treatment of Fabry's Disease with the Pharmacologic Chaperone Migalastat. N Engl J Med. 2016 Aug 11;375(6):545-55. doi: 10.1056/NEJMoa1510198. PMID 27509102

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During Stage 1 (0-6 Months), all participants were randomized to either Migalastat or Placebo. After Stage 1, all participants progressed to Stage 2 where they received open-label migalastat for 6 months (>6-12 Months). After Stage 2, participants were eligible to enter the optional, 12-month, open-label extension (OLE) (>12-24 Months).
Groups:
- Migalastat (0-6 Months): Migalastat hydrochloride (migalastat) 150-milligram (mg) capsule (equivalent to 123 mg of migalastat) given orally every other day (QOD) during the 6-month, double-blind, randomized placebo-controlled treatment period (Stage 1). After Stage 1, participants progressed to Stage 2 where they received open-label migalastat for 6 months.
- Placebo (0-6 Months): Placebo capsule given orally QOD during the 6-month, double-blind, randomized placebo-controlled treatment period (Stage 1). After Stage 1, participants progressed to Stage 2 where they received open-label migalastat for 6 months.
- Migalastat (>6-12 Months): Migalastat 150-mg capsule given orally QOD during the 6-month open-label treatment period (Stage 2). Includes all participants who progressed from both the migalastat (0-6 Months) and the placebo (0-6 Months) Stage 1 treatment groups. After Stage 2, participants were eligible to enter the optional, 12-month OLE.
- Migalastat (>12-24 Months): Migalastat 150-mg capsule given orally QOD for up to 12 months during the optional OLE. Includes all participants who decided to continue treatment after completing the 6-month, open-label Stage 2 treatment period.
Period: 6-Month Double-blind (Stage 1)
Arm/Group | Migalastat (0-6 Months) | Placebo (0-6 Months) | Migalastat (>6-12 Months) | Migalastat (>12-24 Months)
Started | 34 | 33 | 0 (Zero participants noted because participants did not start Stage 2 yet.) | 0 (Zero participants noted because participants did not start the OLE yet.)
Received at Least 1 Dose of Study Drug | 34 | 33 | 0 | 0
Intent-to-Treat (ITT) (All randomized participants regardless of their participation in the study beyond Randomization.) | 34 | 33 | 0 | 0
Modified Intent-to-Treat (mITT) (Participants with Baseline and Month 6 biopsy results.) | 30 | 30 | 0 | 0
Completed | 34 | 30 | 0 | 0
Not Completed | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Period: 6-Month Open-label (Stage 2)
Arm/Group | Migalastat (0-6 Months) | Placebo (0-6 Months) | Migalastat (>6-12 Months) | Migalastat (>12-24 Months)
Started | 0 (Zero participants noted because participants had completed Stage 1.) | 0 (Zero participants noted because participants had completed Stage 1.) | 63 (One participant (Migalastat [0-6 Months]) withdrew consent after completing Month 6.) | 0 (Zero participants noted because participants did not start the OLE yet.)
ITT-amenable (Amenable mutations based on Good Laboratory Practice (GLP) Human Embryonic Kidney (HEK) assay.) | 0 | 0 | 47 | 0
Completed | 0 | 0 | 60 | 0
Not Completed | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Period: 12-Month Open-label Extension (Optional)
Arm/Group | Migalastat (0-6 Months) | Placebo (0-6 Months) | Migalastat (>6-12 Months) | Migalastat (>12-24 Months)
Started | 0 (Zero participants noted because participants had completed Stage 1.) | 0 (Zero participants noted because participants had completed Stage 1.) | 0 (Zero participants noted because participants had completed Stage 2.) | 57 (The OLE was optional for those who completed Stage 2. Reasons for not entering were not recorded.)
ITT-amenable (Amenable mutations based on GLP HEK assay.) | 0 | 0 | 0 | 42
Completed | 0 | 0 | 0 | 54
Not Completed | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Migalastat-Migalastat: Migalastat 150-mg capsule given orally QOD during the 6-month, double-blind, randomized placebo-controlled treatment period (Stage 1), during the 6-month open-label treatment period (Stage 2), and for up to 12 months during the OLE.
- Placebo-Migalastat: Placebo capsule given orally QOD during the 6-month, double-blind, randomized placebo-controlled treatment period (Stage 1). Migalastat 150-mg capsule given orally QOD during the 6-month open-label treatment period (Stage 2) and for up to 12 months during the OLE.
- Total: Total of all reporting groups
Arm/Group | Migalastat-Migalastat | Placebo-Migalastat | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (13.29) | 44.5 (10.18) | 42.2 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants With At Least A 50% Reduction From Baseline To Month 6 In The Average Number Of Kidney Interstitial Capillary (IC) Globotriaosylceramide (GL-3) Inclusions
Description: Renal biopsies were taken at Baseline and Month 6 (Stage 1). The specimens were evaluated using virtual microscopy. The annotation, scoring, and adjudication of the kidney histology assessments were performed by the Clinical Pathology Endpoints Committee. The number of kidney IC GL-3 inclusions was assessed by 3 renal pathologists who were blinded to treatment assignments, participants' data, and biopsy sequence. One pathologist served as annotator and identified the 300 capillaries on up to 8 slides per specimen to be scored. Two pathologists served as scorers; these pathologists completed the blinded paired assessments. Each pathologist served as annotator/adjudicator for 1/3 of the cases. Paired assessments were undertaken at Baseline and Month 6. Assessments were made using digital images. A responder was defined as a participant with a ≥50% reduction from Baseline to Month 6 in the average number of kidney IC GL-3 inclusions.
Time Frame: Baseline, Month 6
Population: ITT: All randomized participants regardless of their participation in the study beyond randomization. As per the statistical analysis plan, analysis excluded participants who were missing baseline kidney biopsy results.
Measure: Count of Participants; unit: Participants
Groups:
- Migalastat: Migalastat 150-mg capsule given orally QOD during the 6-month, double-blind, randomized placebo-controlled treatment period (Stage 1).
- Placebo: Placebo capsule given orally QOD during the 6-month, double-blind, randomized placebo-controlled treatment period (Stage 1).
Arm/Group | Migalastat | Placebo
Number analyzed (Participants) | 32 | 32
Participants
  Responder | 13 | 9
  Non-Responder | 19 | 23
Statistical Analysis 1: Comparison: Migalastat vs Placebo; Test type: Superiority; p = 0.2996, Cochran-Mantel-Haenszel; p-value from Cochran-Mantel-Haenszel test stratified by sex; Difference = 12.5, 95% CI 2-sided [-13.4 to 37.3] — The difference between the percentage of successes between migalastat and placebo treatment groups

2. Secondary Outcome: Percent Change In Kidney IC GL-3 Inclusions From Baseline To Month 6
Description: Renal biopsies were taken at Baseline and Month 6. The specimens were evaluated using virtual microscopy. The annotation, scoring, and adjudication of the kidney histology assessments were performed by the Clinical Pathology Endpoints Committee. The number of kidney IC GL-3 inclusions was assessed by 3 renal pathologists who were blinded to treatment assignments, participants' data, and biopsy sequence. One pathologist served as annotator and identified the 300 capillaries on up to 8 slides per specimen to be scored. Two pathologists served as scorers; these pathologists completed the blinded paired assessments. Each pathologist served as annotator/adjudicator for 1/3 of the cases. Paired assessments were undertaken at Baseline and Month 6. Assessments were made using digital images.
Time Frame: Baseline, Month 6
Population: ITT: All randomized participants regardless of their participation in the study beyond randomization.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Migalastat | Placebo
Number analyzed (Participants) | 34 | 33
percent change | -7.948 (105.2736) | 12.985 (90.5131)

3. Secondary Outcome: Change From Baseline Through Month 24 In Urine GL-3 Levels
Description: The effect of migalastat versus placebo on urine GL-3 levels was measured by liquid chromatography-mass spectrometry/mass spectrometry. The 24-hour urine samples were collected at Baseline, Month 6 (Stage 1), Month 12 (Stage 2), and Month 24 (OLE). Results are presented as changes in nanograms (ng)/mg creatinine from Baseline to the end of the 3 stages.
Time Frame: Baseline, Months 6, 12, and 24
Population: Stage 1: ITT, all randomized participants regardless of participation in the study beyond randomization. Stage 2: participants who completed Stage 1 and entered Stage 2. OLE: participants who completed Stage 2 and entered the optional OLE. Once assay and sample issues were identified, later samples were not further analyzed; all data was listed.
Measure: Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Migalastat-Migalastat | Placebo-Migalastat
Number analyzed (Participants) | 33 | 30
ng/mg creatinine
  Stage 1 | -234.80 (853.451) | -186.24 (957.119)
  Stage 2: number analyzed (Participants) | 31 | 28
  Stage 2 | -179.63 (699.157) | -537.95 (1169.883)
  OLE: number analyzed (Participants) | 12 | 9
  OLE | -62.37 (615.944) | -177.42 (288.224)

4. Other Pre Specified Outcome: Change From Month 6 To Month 12 In Average Number Of Kidney IC GL-3 Inclusions
Description: Renal biopsies were taken at Month 6 and Month 12. The specimens were evaluated using virtual microscopy. The annotation, scoring, and adjudication of the kidney histology assessments were performed by the Clinical Pathology Endpoints Committee. The number of kidney IC GL-3 inclusions was assessed by 3 renal pathologists who were blinded to treatment assignments, participants' data, and biopsy sequence. One pathologist served as annotator and identified the 300 capillaries on up to 8 slides per specimen to be scored. Two pathologists served as scorers; these pathologists completed the blinded paired assessments. Each pathologist served as annotator/adjudicator for 1/3 of the cases. Paired assessments were undertaken at Month 6 and Month 12. Assessments were made using digital images.
Time Frame: Month 6, Month 12
Population: mITT with amenable mutations: Randomized participants who switched from placebo to migalastat during Stage 2, received at least 1 dose of study drug, and underwent a renal biopsy at both Baseline and Month 6. Amenable mutations are mutant forms of α-galactosidase A (α Gal-A) amenable to migalastat. Amenable mutations based on the GLP HEK assay.
Measure: Least Squares Mean (95% Confidence Interval); unit: kidney IC GL-3 inclusions
Groups:
- Placebo-Migalastat: Placebo capsule given orally QOD during the 6-month, double-blind, randomized placebo-controlled treatment period (Stage 1). Migalastat 150-mg capsule given orally QOD during the 6-month open-label treatment period (Stage 2).
Arm/Group | Placebo-Migalastat
Number analyzed (Participants) | 20
kidney IC GL-3 inclusions | -0.320 [-0.5719 to -0.0677]
Statistical Analysis 1: Comparison: Placebo-Migalastat; Test type: Other — Mixed effects model for repeated measures (MMRM) approach with fixed effects of treatment, time (Month 6 and Month 12), mutation type (amenable or non-amenable), time by treatment interaction, time by mutation type interaction, and the baseline value as a covariate. An unstructured covariance matrix to account for repeated measures within a participant was assumed; p = 0.014, MMRM — Significant at the 0.050 level

5. Post Hoc Outcome: Change From Baseline To Month 6 In Average Number Of Kidney IC GL-3 Inclusions
Description: Renal biopsies were taken at Baseline and Month 6. The specimens were evaluated using virtual microscopy. The annotation, scoring, and adjudication of the kidney histology assessments were performed by the Clinical Pathology Endpoints Committee. The number of kidney IC GL-3 inclusions was assessed by 3 renal pathologists who were blinded to treatment assignments, participants' data, and biopsy sequence. One pathologist served as annotator and identified the 300 capillaries on up to 8 slides per specimen to be scored. Two pathologists served as scorers; these pathologists completed the blinded paired assessments. Each pathologist served as annotator/adjudicator for 1/3 of the cases. Paired assessments were undertaken at Baseline and Month 6. Assessments were made using digital images. Treatment effect was estimated using the LS mean difference between treatments within the context of the ANCOVA model.
Time Frame: Baseline, Month 6
Population: ITT-amenable: Randomized participants with amenable mutations who received study drug during Stage 1. Amenable mutations are mutant forms of α Gal-A amenable to migalastat. Amenable mutations based on the GLP HEK assay. Participants were analyzed according to their original randomized treatment group.
Measure: Mean (Standard Deviation); unit: kidney IC GL-3 inclusions
Arm/Group | Migalastat
Number analyzed (Participants) | 25
kidney IC GL-3 inclusions | -0.250 (0.5126)
Statistical Analysis 1: Comparison: Migalastat; The change from Baseline in the average number of kidney ICs was analyzed using an ANCOVA model with covariate adjustment for the baseline value and factors for treatment group and the treatment by baseline interaction; Test type: Other; p = 0.0078, ANCOVA — Significant at the 0.010 level; Difference LSMeans = -0.3, 95% CI 2-sided [-0.6 to -0.1]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were monitored up to 25 months (±7 days) after the first dose of study drug. AEs were reported from the first dose of study medication at Baseline (Visit 1) in Stage 1 to 1 month (±7 days) after the date of the last study visit, whether during Stage 1, Stage 2, or the optional OLE, or after premature discontinuation from the study.
Description: Stage 1 AEs were any AEs that started between the first dose of Stage 1 and the first dose of Stage 2 (or last Stage 1 administration for participants that discontinued during Stage 1). Stage 2 AEs were any AEs that started between the first dose of Stage 2 and the first dose of the OLE (or the last Stage 2 administration for participants that discontinued during Stage 2). OLE AEs were any AEs that started after the first dose of the OLE.
Groups:
- Migalastat (0-6 Months): Migalastat 150-mg capsule given orally QOD during the 6-month, double-blind, randomized placebo-controlled treatment period (Stage 1). After Stage 1, participants progressed to Stage 2 where they received open-label migalastat for 6 months.
- All Migalastat (>6-12 Months): Migalastat 150-mg capsule given orally QOD during the 6-month open-label treatment period (Stage 2). Includes all participants who progressed from both the migalastat (0-6 Months) and the placebo (0-6 Months) Stage 1 treatment groups. After Stage 2, participants were eligible to enter the optional, 12-month OLE.
- All Migalastat (>12-24 Months): Migalastat 150-mg capsule given orally QOD for up to 12 months during the optional OLE. Includes all participants who decided to continue treatment after completing the 6-month, open-label Stage 2 treatment period.
Arm/Group | Migalastat (0-6 Months) | Placebo (0-6 Months) | All Migalastat (>6-12 Months) | All Migalastat (>12-24 Months)
Serious Adverse Events (participants affected / at risk) | 2/34 | 4/33 | 5/63 | 11/57
Other Adverse Events (participants affected / at risk) | 31/34 | 30/33 | 50/63 | 46/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat (0-6 Months) (N=34) | Placebo (0-6 Months) (N=33) | All Migalastat (>6-12 Months) (N=63) | All Migalastat (>12-24 Months) (N=57)
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anaplastic Large Cell Lymphoma T - and Null - Cell Types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Bulimia Nervosa (Psychiatric disorders) | 0 | 0 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bone Cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bacterial Infection (Infections and infestations) | 0 | 1 | 0 | 0
Helicobacter Gastritis (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis Viral (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat (0-6 Months) (N=34) | Placebo (0-6 Months) (N=33) | All Migalastat (>6-12 Months) (N=63) | All Migalastat (>12-24 Months) (N=57)
Fatigue (General disorders) | 4 | 4 | 2 | 3
Pyrexia (General disorders) | 4 | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 3 | 4
Insomnia (Psychiatric disorders) | 3 | 2 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 1 | 7 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 1
Paraesthesia (Nervous system disorders) | 4 | 4 | 4 | 2
Headache (Nervous system disorders) | 12 | 7 | 9 | 6
Vertigo (Ear and labyrinth disorders) | 2 | 3 | 3 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 2
Dry Mouth (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 5 | 2
Nausea (Gastrointestinal disorders) | 4 | 2 | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 3
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 9
Haematuria (Renal and urinary disorders) | 3 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 5
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 6
Influenza (Infections and infestations) | 0 | 3 | 0 | 2
Nasopharyngitis (Infections and infestations) | 6 | 2 | 5 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 3 | 5 | 3
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 3 | 5
Atrial Fibrillation (Cardiac disorders) | 2 | 0 | 1 | 3
Abdominal Distension (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Asthenia (General disorders) | 2 | 1 | 0 | 1
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Weight Increased (Investigations) | 2 | 1 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 2 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 3

LIMITATIONS AND CAVEATS:
During Phase 3, prior to unblinding, the assay used for enrollment was validated (GLP HEK assay). Mutant forms of α-Gal A that met assay criteria were categorized as amenable; additional analyses were subsequently performed on this target population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only the results from this trial, provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review prior to submission for publication. If requested and prior to publication, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.